CLINICAL TRIAL: NCT05149391
Title: A Phase 1 Study of CD19 and CD20 Targeted Chimeric Antigen Receptor T Cells Therapy (C-CAR039) in Subjects With Relapsed and/or Refractory B Cell Non-Hodgkin's Lymphoma
Brief Title: A Study of C-CAR039 in Subjects With Relapsed and/or Refractory B Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Zhu, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0702-022
Record Dates: First submitted 2021-11-09; First posted 2021-12-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2021-11

CONDITIONS: B Cell Non-Hodgkin's Lymphoma
Keywords: CD19/CD20-directed Chimeric Antigen Receptor T Cells
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-CAR039 (Experimental): Autologous C-CAR039 administered by intravenous (IV) infusion
  Interventions: Biological: CD19/CD20-directed Chimeric Antigen Receptor T Cells

INTERVENTIONS:
Biological: CD19/CD20-directed Chimeric Antigen Receptor T Cells — Autologous 2nd generation CD19/CD20-directed Chimeric Antigen Receptor T Cells, single infusion intravenously
  Other Names: C-CAR039

SUMMARY:
This is a single-center, open-label study to evaluate the safety and efficacy of C-CAR039 in relapsed and/or refractory B cell Non-Hodgkin's Lymphoma patients.

DETAILED DESCRIPTION:
The study includes the following sequential phases: Screening, Apheresis and C-CAR039 manufacturing, Baseline testing, Lymphodepletion, C-CAR039 infusion, Dose-limiting toxicity observation and Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study and signed the Informed Consent;
2. Age, 18-70 years (include 18 and 70), male or female;
3. Expected survival ≥ 12 weeks
4. Eastern Cooperative Oncology Group score 0-2
5. CD19 or CD20 positive B-Non-Hodgkin's lymphoma confirmed by cytology or histology according to World Health Organization 2016 criteria;
6. Patients with a clear diagnosis of relapsed and/or refractory B-Non-Hodgkin's lymphoma, including Diffuse Large B Cell Lymphoma, Follicular Lymphoma and Mantle Cell Lymphoma. Diffuse Large B Cell Lymphoma includes the following types:

   1. Diffuse Large B Cell Lymphoma, Non Specifically
   2. Primary Mediastinal B-cell Lymphoma
   3. Transformed Follicular Lymphoma
   4. High Grade B-Cell Lymphoma With MYC and BCL2 and/or BCL6
   5. High Grade B-Cell Lymphoma, Non Specifically
7. For CD20-positive subjects, they should have received at least one regimen containing anti-CD20-targeted therapy (such as rituximab). If they do not complete the regimen due to intolerance, the cause of intolerance should be recorded;
8. No contraindications of apheresis.
9. At least one measurable lesion according to Lugano 2014 criteria;
10. Adequate organ function and adequate bone marrow reserve

    1. Hemoglobin≥80 g/L
    2. Absolute neutrophil count≥1.0×109/L
    3. Platelet≥50×109/L,
    4. Creatinine≤1.5×upper limit of the normal range (ULN)
    5. Cardiac ejection fraction≥50%
    6. Saturation of Pulse Oxygen>92%
    7. Total bilirubin≤1.5×ULN
    8. Alanine Aminotransferase/Aspartate Aminotransferase≤3×ULN

Exclusion Criteria:

1. Malignant tumors other than B-Non-Hodgkin's lymphoma within 5 years prior to screening, except cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and breast ductal carcinoma in situ after radical surgery;
2. Human Immunodeficiency Virus, Hepatitis B Virus, Hepatitis C Virus or treponema pallidum infection ;
3. Any instability of systemic disease, including but not limited to active infection (except local infection), severe cardiac, liver, kidney, or metabolic disease need treatment;
4. Female subjects who have been pregnant or breastfeeding, or who plan to conceive during or within 1 year after treatment, or male subjects' partner plans to conceive within 1 year after their cell transfusion;
5. Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment;
6. Patients who have been previously infected with tuberculosis;
7. Administered Corticosteroids and/or other immunosuppressants within 7 days before apheresis. and 5 days before the infusion of C-CAR039;
8. Patients with central nervous system involvement;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Safety Observation | up to 24 Months. Incidence and severity of adverse events after C-CAR039 infusion according to National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 criteria, including dose-limiting toxicity (DLT) and laboratory abnormalities.
  Incidence of adverse events after C-CAR039 infusion. Incidence and severity of adverse events according to NCI-CTCAE v5.0 criteria, including Dose Limited Toxicity

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of C-CAR039 in the peripheral blood. | Baseline, Days 4, 7, 10 and weeks 2, 3, 4, 8, 12 and month 6, 9, 12, 15, 18, 21, 24
  Detect Chimeric Antigen Receptor-T copies number by quantitative polymerase chain reaction(qPCR).
Time to maximum concentration (Tmax) of C-CAR039 in the peripheral blood. | Baseline, Days 4, 7, 10 and weeks 2, 3, 4, 8, 12 and month 6, 9, 12, 15, 18, 21, 24
  Detect Chimeric Antigen Receptor-T copies number by qPCR.
Peripheral blood duration of C-CAR039 in the peripheral blood after infusion. | Baseline, Days 4, 7, 10 and weeks 2, 3, 4, 8, 12 and month 6, 9, 12, 15, 18, 21, 24
  Detect Chimeric Antigen Receptor-T copies number by qPCR.
Area under the curve 0h-28d of C-CAR039 in the peripheral blood. | Baseline, Days 4, 7, 10 and weeks 2, 3, 4
  Detect Chimeric Antigen Receptor-T copies number by qPCR.
Overall response rate (ORR) | 4 weeks, 12 weeks, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  Complete response (CR) rate plus partial response (PR) rate by Lugano 2014 criteria.
Duration of response (DOR) | up to 24 months
  The time from the date of first response (PR or better) to the date of disease progression or death after C-CAR039 infusion.
Progression-free survival (PFS) | 4 weeks, 12 weeks, 6 months, 9 months, 12 months, 15 months, 18 months, 21 months, 24 months
  The time from C-CAR039 infusion to the date of progression as assessed by Lugano 2014 criteria or death.
Overall survival (OS) | up to 24 months
  The time from C-CAR039 infusion to the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No